CLINICAL TRIAL: NCT04495491
Title: Prediction of the Degree of Angle Opening Distance in Patients With Primary Angle Closure Suspect After Laser Peripheral Iridotomy
Brief Title: Predicting the Effect of Laser Peripheral Iridotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Mingkai Lin, chief physician, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2019KYPJ182
Record Dates: First submitted 2020-07-22; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Glaucoma
Keywords: laser peripheral iridotomy; primary angle closure suspect; angle closure mechanism
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pupillary block group: According to the configurations of angle closure, the pupillary block group is defined as the iris bombe.
  Interventions: Other: pupillary block group
- plateau iris group: According to the configurations of angle closure, the plateau iris group is defined as the thickness of the peripheral iris.
  Interventions: Other: plateau iris group
- mixed mechanism group: According to the configurations of angle closure, the mixing mechanism group is defined as the iris bombe plus thickening of the peripheral iris.
  Interventions: Other: mixing mechanism group

INTERVENTIONS:
Other: pupillary block group — According to the configurations of angle closure, the pupillary block group is defined as the iris bombe.
  Groups: Pupillary block group
Other: plateau iris group — According to the configurations of angle closure, the plateau iris group is defined as the thickness of the peripheral iris.
  Groups: plateau iris group
Other: mixing mechanism group — According to the configurations of angle closure, the mixing mechanism group is defined as the iris bombe plus thickening of the peripheral iris.
  Groups: mixed mechanism group

SUMMARY:
This study will compare the angle parameters of patients with PACS before and after LPI. The investigators will analyze the results of patients with different angle closure mechanisms before and after LPI, and participants hope to find the structural parameters for predicting the effect of LPI.

DETAILED DESCRIPTION:
Primary angle-closure glaucoma is the leading cause of blindness worldwide. It is associated with increased intraocular pressure, which causes optic nerve damage and field defects if untreated. The aqueous humor leaves the anterior chamber through the trabecular meshwork and flows into the aqueous vein and the superior scleral vein through the collector channels and Schlemm's canal. If the trabecular meshwork is not blocked, a wide angle allows enough aqueous humor to drain out. The iris corneal translocation may lead to angle-closure glaucoma.

Laser peripheral iridectomy is recognized as the best surgical method to relieve pupil block. Previous studies have shown increased anterior chamber depth (ACD), area (ACA), and volume (ACV), and increased Angle open distance (AOD) after LPI surgery.

However, postoperative outcomes of LPI were not the same for patients with different angle closure mechanisms.

Postoperative outcomes for LPI were best for patients with pupillary block type, but were moderate for patients with plateau iris group and mixed group.

The purpose of this study, conducted in Chinese subjects, aims to use UBM to evaluate changes in the anterior segment parameters of LPI, and to propose methods to predict postoperative outcomes of LPI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was diagnosed of primary angle closure angle suspect;
2. received ultrasound Biomicroscopy before and after laser peripheral iridotomy;
3. Voluntary participation in this study;
4. Have enough language comprehension ability;
5. Patient or his legal representative has sign the informed consent.

Exclusion Criteria:

1. severe health problems resulting in a life expectancy of less than 1 year;
2. previous intraocular surgery or penetrating eye injury;
3. media opacity preventing laser peripheral iridotomy;
4. Researchers think not suitable to participate in this clinical trial subjects;
5. Refused to sign the informed consent.;
6. There are important viscera function failure or other serious disease, including clinical related coronary artery disease, cardiovascular disease or myocardial infarction into the group of the first six months; serious neurological or psychiatric illness; serious infections; coagulant function abnormality; general active infectious diseases; malignant tumor; serious immune diseases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Patient was diagnosed of primary angle closure angle suspect
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
the changes in anterior opening distance before and after LPI | between the baseline and 1 hour before discharge
  To compare the difference of anterior opening distance after LPI and baseline parameters before LPI. Anterior opening distance, measured on a line perpendicular to the plane of the trabecular surface 500 μm anterior to the scleral spur and extended to meet the surface of the iris

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Lin, MD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-San University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-San Univerdity, Guangzhou, Guangdong, China

REFERENCES:
- [Background] He M, Jiang Y, Huang S, Chang DS, Munoz B, Aung T, Foster PJ, Friedman DS. Laser peripheral iridotomy for the prevention of angle closure: a single-centre, randomised controlled trial. Lancet. 2019 Apr 20;393(10181):1609-1618. doi: 10.1016/S0140-6736(18)32607-2. Epub 2019 Mar 14. PMID 30878226
- [Background] He M, Friedman DS, Ge J, Huang W, Jin C, Lee PS, Khaw PT, Foster PJ. Laser peripheral iridotomy in primary angle-closure suspects: biometric and gonioscopic outcomes: the Liwan Eye Study. Ophthalmology. 2007 Mar;114(3):494-500. doi: 10.1016/j.ophtha.2006.06.053. Epub 2006 Nov 21. PMID 17123610
- [Background] He M, Foster PJ, Ge J, Huang W, Zheng Y, Friedman DS, Lee PS, Khaw PT. Prevalence and clinical characteristics of glaucoma in adult Chinese: a population-based study in Liwan District, Guangzhou. Invest Ophthalmol Vis Sci. 2006 Jul;47(7):2782-8. doi: 10.1167/iovs.06-0051. PMID 16799014